CLINICAL TRIAL: NCT00263783
Title: Phase I Trial of Weekly MEDI-522 in Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Luz Hammershaimb, M.D., V.P., Clinical Dev., MedImmune Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP065
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — etaracizumab

ARMS (1):
- 1 (Experimental): MEDI-522
  Interventions: Drug: MEDI-522

INTERVENTIONS:
Drug: MEDI-522 — MEDI-522 will be administered at doses of 1.0, 2.0, 4.0, 6.0, 8.0, and 10.0 mg/kg. [As a 30 minute IV infusion initially as a single dose (single-dose treatment period) and 2 to 5 weeks later as weekly doses (multiple-dose treatment period) for up to 1 year.]

SUMMARY:
To determine the safety profile of single and multiple doses of MEDI522 in patients with refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or post menopausal female patients with histologically confirmed advanced refractory solid tumors for which no reasonable therapy exists. Patient is not required to have measurable disease.
* Age >18 years
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (see APPENDIX 1 for details).
* Patients who had prior surgery, radiation, or chemotherapy will be eligible provided at least 4 weeks have elapsed prior to study initiation. Patients must have recovered from treatment-related toxicities, and surgical wounds must be healed.
* Patients who have had prior immunotherapy with approved agents are eligible.
* Patients must have hemoglobin >10.0 g/dL, ANC >1,000/mm3, WBC >3,000/mm3,000/mm3, platelets ³100,000/mm3, bilirubin £2.0 mg/dL, AST/ALT no greater than 5 times the upper limit of normal (ULN), and serum creatinine <1.5 mg/dL (or calculated creatinine clearance ³60 mL/min).
* Patients must have prothrombin time (PT) and partial thromboplatin time (PTT) less than upper limit of normal or international normalized ratio (INR) less than 1.1.
* Patients must have thyroxine (T4) and thyroid-stimulating hormone (TSH) within normal limits.
* Patients must be informed of and understand the investigational nature of this trial and give written informed consent prior to receipt of any study medication or beginning study procedures.

Exclusion Criteria:

* Patient has known brain metastases or primary brain tumors, symptomatic pleural effusion or ascites requiring paracentesis.
* Patient has respiratory insufficiency requiring oxygen treatment, or has lymphangitic involvement of lungs.
* Patient has evidence of hematemesis, melena, hematochezia, or hematuria (2 or greater on urine dipstick).
* Patient has a history of a significant adverse event related to previously administered humanized monoclonal antibody.
* Patient has known HIV or hepatitis virus infection.
* Patient has prior myocardial infarction or angina, or uncontrolled hypertension (systolic BP >140 mm Hg).
* Patient has either prior strokes or transient ischemic attacks.
* Patient has active infections requiring systemic antiinfective therapy or other physical or psychological illnesses that would preclude drug administration or patient compliance.
* Patient has donated blood or received an investigational agent in the last 4 weeks.
* Patient has a history of active illness or behavior, including substance dependence or abuse that, in the opinion of the investigator, might pose additional risk in administering the study drug to the patient.
* General medical or psychological conditions that would not permit the patient to complete the study or sign the informed consent

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2001-03; Primary Completion 2002-04 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Safety: The incidence and severity of adverse experiences and laboratory abnormalities will be tabulated and presented overall and by dose. | Study Day 1 up to 8 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Will be assessed using the variables of area under the concentration curve (AUC) which will be calculated by the trapezoidal rule, peak concentration (Cmax), time to peak concentration (Tmax), half life | 35 days after the first dose
Measured pharmacokinetic parameters may be one of the factors used in determination of the Phase II regimen. | Appx. 5 days after the 4th weekly dose
Antitumor Activity: The antitumor activity of MEDI-522 in patients with refractory solid tumors will be assessed by calculating tumor response rate and time to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Luz Hammershaimb, MD, Study Director — MedImmune LLC
Locations (1):
- Institut Gustave Roussy, Villejuf, France